CLINICAL TRIAL: NCT01778660
Title: Standard Versus Mnemonic Counseling for Fecal Incontinence: a Pilot Randomised Control Trial
Brief Title: Standard Versus Mnemonic Counseling for Fecal Incontinence
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Sara Cichowski, Principal Investigator, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTSC-12-429; CTSTC025-3 (Other: CTSC)
Record Dates: First submitted 2013-01-16; First posted 2013-01-29 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2013-01

CONDITIONS: Fecal Incontinence; Counselling; Patient Satisfaction
Keywords: Fecal Incontinence; Treatment options; Patient Satisfaction
MeSH Terms: conditions — Fecal Incontinence; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Counselling (Active Comparator): Patients in this arm are randomised to standard counselling.
  Interventions: Other: Standard
- Mnemonic Counselling (Experimental): Patients in this arm are randomised to counselling with the aid of a mnemonic.
  Interventions: Other: Type of Counselling (Mnemonic)

INTERVENTIONS:
Other: Type of Counselling (Mnemonic)
  Arms: Mnemonic Counselling
Other: Standard
  Arms: Standard Counselling

SUMMARY:
This study compares standard versus mnemonic counseling for the treatment of fecal incontinence. A mnemonic is a word or rhyme used to aid memory. Our hypothesis is that women randomised to mnemonic counseling will higher recall of treatments, satisfaction with the physician visit and greater improvement in their quality of life when compared to women who received standard counseling.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosed with fecal incontinence by on of the attending physicians
* Bothersome fecal incontinence symptoms for at least 3 months
* Able to give informed consent
* Able to speak, read and comprehend English

Exclusion Criteria:

* Younger than 18 years
* Fecal Incontinence <3 months
* Unable to give informed consent
* Unable to speak, read and comprehend English
* Diagnosis of active colorectal or anal malignancy, inflammatory bowel disease, recto-vaginal fistula, and rectal prolapse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Recall | We are measuring the difference in recall the day of the physician counseling and 2 months after physician counselling
  Patients will be asked to recall treatments recommended for fecal incontinence.

SECONDARY OUTCOMES:
Questionare on the Quality of the Physician and Patient Interaction | Patients will complete this questionnaire following the physician counseling on day 1 of enrollment.
Modified Manchester | We are comparing the score change from after the physician counselling on day 1 of enrollment and at 2 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cichowski, M.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Cichowski SB, Dunivan GC, Rogers RG, Murrietta AM, Komesu YM. Standard compared with mnemonic counseling for fecal incontinence: a randomized controlled trial. Obstet Gynecol. 2015 May;125(5):1063-1070. doi: 10.1097/AOG.0000000000000755. PMID 25932833